CLINICAL TRIAL: NCT03259425
Title: Phase II Neoadjuvant Trial of Nivolumab in Combination With HF10 Oncolytic Viral Therapy in Resectable Stage IIIB, IIIC, IVM1a Melanoma (Neo-NivoHF10)
Brief Title: Neoadjuvant Trial of Nivolumab in Combination With HF10 Oncolytic Viral Therapy in Resectable Stage IIIB, IIIC, IVM1a Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DSMC Recommendation
Sponsor: University of Utah (Other)
Collaborators: Bristol-Myers Squibb (Industry); Takara Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI102346
Record Dates: First submitted 2017-08-18; First posted 2017-08-23 (Actual); Results first posted 2019-10-10 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Melanoma
Keywords: Resectable Stage IIIB, IIIC, and IVM1a
MeSH Terms: conditions — Melanoma | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: This is a single-arm, open label, Phase II
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nivolumab and HF10, all participants (Experimental)
  Interventions: Drug: Nivolumab; Drug: HF10

INTERVENTIONS:
Drug: Nivolumab — Nivolumab at a dose of 240 mg given as an IV infusion starting on day 0. It will be given every 14 days for a total of 7 infusions; Then participant will undergo surgery. Nivolumab will then be administered at a flat dose of 480 mg IV every 28 days for up to one year.
  Other Names: OPDIVO
Drug: HF10 — 1 x 107th TCID50/mL, intratumoral injection to a single or multiple eligible tumors for a total of 5 mL; on days 0, 7, 14, 21, 28, 42, 56, 70, 84 for a total of 9 injections. All eligible tumors except one will be treated with HF10 up to the maximum volume allowed. The untreated tumor will be used as an untreated control lesion.

SUMMARY:
This is a single-arm, open label, Phase II study evaluating the safety and efficacy of neoadjuvant Nivolumab and HF10 in resectable stage IIIB, IIIC, and IVM1a melanoma.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be >18 years or older.
* Participants must have stage IIIB, IIIC, or IVM1a (equivalent staging at time of enrollment via American Joint Committee on Cancer (AJCC) 7th edition) metastatic melanoma which is eligible for complete surgical resection.
* Prior systemic, regional and radiation anticancer therapies must have been completed at least three months prior to enrollment. Prior therapies (including anti-programmed death (PD)-1 inhibitors) are allowed provided three months have elapsed from last dose.
* Participants must be a candidate for intralesional therapy.
* At least 1 injectable cutaneous, subcutaneous, or nodal melanoma lesion > 10 mm in longest diameter OR
* Multiple injectable melanoma lesions which in aggregate have a longest diameter of > 10 mm AND
* Must have no known bleeding diathesis or coagulopathy that would make intratumoral injection unsafe.
* Participants must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Serum (LDH) level < 1.5 upper limit of normal (ULN) within 28 days prior to enrollment.
* Participants have adequate organ function within 28 days prior to enrollment, as defined in the protocol
* Men and women of childbearing potential must agree to use adequate contraception from the time of consent through 7 months after final nivolumab study treatment.
* Females of childbearing potential must have a negative urine or serum pregnancy test within 1 week prior to the start of treatment.
* Participants must be able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.

Exclusion Criteria:

* Participants with active visceral, central nervous system, or any bone metastases melanoma (Stage IVM1b or IVM1c).
* Participants whose primary diagnosis was ocular melanoma.
* Participants receiving anti-herpes medication (i.e., acyclovir, famciclovir, or valacyclovir) within 1 week prior to initiating HF10 treatment. Participants may not require intermittent or chronic systemic (intravenous or oral) treatment with an antiherpetic drug other than intermittent topical use.
* Participants who have an active herpetic skin lesion(s) or prior complications of herpes simplex virus (HSV)-1 infection.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, as determined by the investigator.
* Medical history of autoimmune disease (e.g. Crohn's disease, ulcerative colitis) or other disease requiring systemic glucocorticoid or immunosuppressive therapy. Subjects who receive daily steroid replacement therapy serve as an exception to this rule. Daily prednisone equivalent at doses up to 10 mg would qualify.
* Participants with clinically evident Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV), or Epstein-Barr Virus (EBV) infection are excluded.
* Pregnant or breast feeding women; women desiring to become pregnant within the timeframe of the study are also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-09-21 (Actual); Study Completion 2020-09-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Huntsman Cancer Institute, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab and HF10 (All Participants): Nivolumab: Nivolumab at a dose of 240 mg given as an IV infusion starting on day 0. It will be given every 14 days for a total of 7 infusions; Then participant will undergo surgery. Nivolumab will then be administered at a flat dose of 480 mg IV every 28 days for up to one year.
  HF10: 1 x 107th TCID50/mL, intratumoral injection to a single or multiple eligible tumors for a total of 5 mL; on days 0, 7, 14, 21, 28, 42, 56, 70, 84 for a total of 9 injections.
Period: Overall Study
Arm/Group | Nivolumab and HF10 (All Participants)
Started | 7
Surgery | 6
Completed | 6
Not Completed | 1
Not completed — Disease progression to an extent that didn't allow surgery | 1

BASELINE CHARACTERISTICS:
Groups:
- Nivolumab and HF10 (All Participants ): Nivolumab: Nivolumab at a dose of 240 mg given as an IV infusion starting on day 0. It will be given every 14 days for a total of 7 infusions; Then participant will undergo surgery. Nivolumab will then be administered at a flat dose of 480 mg IV every 28 days for up to one year.
  HF10: 1 x 107th TCID50/mL, intratumoral injection to a single or multiple eligible tumors for a total of 5 mL; on days 0, 7, 14, 21, 28, 42, 56, 70, 84 for a total of 9 injections.
Arm/Group | Nivolumab and HF10 (All Participants )
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.14 (22.17)
Age, Continuous [Median (Full Range); unit: years] | 71 [18 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Tumor Viability Percentage [Count of Participants; unit: Participants] — Following a pre-treatment biopsy at baseline, a pathologist reviewed the tumor tissue collected and estimated tumor viability, expressed as a percentage of viable tumor from 0-100%. This is reported here as a count of participants with greater than 90% tumor viability at baseline.
  Participants
    Tumor Viability >= 90% | 7
    Tumor Viability < 90% | 0

OUTCOME MEASURES:

1. Primary Outcome: Pathological Response
Description: Following 12 weeks of neoadjuvant treatment with nivolumab and HF10, participants underwent definitive surgery. A percent viable tumor was assessed semi-quantitatively in the definitive surgical resection specimen by estimating the proportion of residual tumor in relation to the total tumor area and reported as percentage viability. A pathologic complete response was defined as no viable residual melanoma cells in the surgical specimen. A major pathologic response was defined as <50% viable tumor cells. A minor pathologic response was defined as 50% or greater viable tumor cells, including specimens that had 100% viability at surgery.
Time Frame: at time of surgery (12 weeks)
Population: One of seven participants had progressive disease while receiving neoadjuvant therapy and did not receive surgical resection and therefore per protocol was not assessed for response.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and HF10 (All Participants)
Number analyzed (Participants) | 6
Participants
  Pathologic Complete Response (0% Tumor Viability) | 5
  Major Pathologic Response (<50% Tumor Viability) | 0
  Minor Pathologic Response (>=50% Tumor Viability) | 1

2. Secondary Outcome: Recurrence-free Survival: Number of Participants With no Disease Recurrence After Surgery
Description: Recurrence after surgery will be assessed by radiologic scans and confirmed by biopsy. Death within the follow-up period is also considered recurrence. This outcome will report the number of participants who were alive and who had no disease recurrence during the follow-up period.
Time Frame: up to 2 years post-surgery (1 year after end of adjuvant nivolumab, which was given for up to 1 year post-surgery)
Population: The participant who did not complete surgery was not followed for post-surgery outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and HF10 (All Participants)
Number analyzed (Participants) | 6
Participants | 2

3. Secondary Outcome: Overall Survival: Number of Participants Alive One Year After Completing Adjuvant Nivolumab
Description: Participants were followed for survival for one year after completion of adjuvant nivolumab. Adjuvant nivolumab was planned for up to one year of adjuvant treatment after surgery. This objective reports the number of participants who were alive one year after the completion of adjuvant nivolumab.
Time Frame: up to 2 years post-surgery (1 year after end of adjuvant nivolumab, which was given for up to 1 year post-surgery)
Population: The participant who did not complete surgery was not followed for post-surgery outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and HF10 (All Participants)
Number analyzed (Participants) | 6
Participants | 5

4. Secondary Outcome: Radiographic Response: Number of Participants Within Each Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 Response Category
Description: Participants were assessed radiographically and clinically prior to study start and prior to surgery. Lesions were measured, and lesions that were at least 10 mm on CT, MRI, caliper, or ruler, or at least 20 mm on x-ray were documented as Target Lesions. Lesions that did not meet criteria to be Target Lesions were documented as Non-Target lesions. Measurements of Target Lesions were summed. Change in Target Lesion measurements was used to determine response by RECIST 1.1 criteria. Complete Response (CR) indicates a disappearance of all lesions. Partial Response (PR) indicates at least 30% decrease in the sum of Target Lesions. Progressive Disease (PD) indicates at least 20% increase in the sum of Target Lesions, or the appearance of one or more new lesions after baseline. Stable Disease (SD) is neither sufficient shrinkage to qualify as PR nor sufficient increase to qualify as PD. Objective was reported as number of participants within each response category.
Time Frame: 12 weeks from baseline to surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and HF10 (All Participants)
Number analyzed (Participants) | 7
Participants
  Complete Response (CR) | 1
  Partial Response (PR) | 0
  Stable Disease (SD) | 3
  Progressive Disease (PD) | 3

5. Secondary Outcome: Number of Participants With Complete Surgical Resection
Description: Participants' surgical samples were assessed by a pathologist after surgery to determine if complete surgical resection was achieved after neo-adjuvant treatment with nivolumab and HF10. R0 indicates a complete surgical resection was achieved and means no residual tumor was detected after after surgery. R1 means microscopic tumor was detected and a complete surgical resection was not achieved.
Time Frame: Within 28 days after Day 84
Population: The participant who did not complete surgery was not followed for post-surgery outcomes.
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and HF10 (All Participants)
Number analyzed (Participants) | 6
Participants
  R0 Complete Surgical Resection | 5
  R1 Incomplete Surgical Resection | 1

6. Secondary Outcome: Number of Participants With Adverse Events Related to HF10 Treatment
Description: Participants were monitored for adverse events (AEs) during treatment with HF10 using CTCAE v4 criteria. AEs were graded as being mild (grade 1), moderate (grade 2), grade 3 (severe), grade 4 (life-threatening), and grade 5 (fatal). Each adverse event was reviewed by a treating investigator for relatedness to study treatment. For this outcome, the number of participants who experienced any AEs that were possible, probably, or definitely related to HF10 treatment are grouped by grade 1-2 and grade 3-5 AEs.
Time Frame: throughout HF10 treatment (up to 84 days)
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and HF10 (All Participants)
Number analyzed (Participants) | 7
Participants
  Participants with G1-2 AEs related to HF10 | 7
  Participants with G3-5 AEs related to HF10 | 1

7. Secondary Outcome: Number of Participants With Adverse Events Related to Nivolumab Treatment
Description: Participants were monitored for adverse events (AEs) during treatment with nivolumab using CTCAE v4 criteria. AEs were graded as being mild (grade 1), moderate (grade 2), grade 3 (severe), grade 4 (life-threatening), and grade 5 (fatal). Each adverse event was reviewed by a treating investigator for relatedness to study treatment. For this outcome, the number of participants who experienced any AEs that were possible, probably, or definitely related to nivolumab treatment are grouped by grade 1-2 and grade 3-5 AEs.
Time Frame: throughout nivolumab treatment (up to 84 days prior to surgery and up to 1 year after surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | Nivolumab and HF10 (All Participants)
Number analyzed (Participants) | 7
Participants
  Participants with G1-2 AEs related to Nivolumab | 7
  Participants with G3-5 AEs related to Nivolumab | 2

ADVERSE EVENTS:
Time Frame: From first dose of study treatment to 30 days after last dose of study treatment (up to 1 year, 8 months)
Description: Per protocol: The occurrence of adverse events should be sought by non-directive questioning of the participant at each visit or phone contact during the study. Adverse events also may be detected when they are volunteered by the participant during or between visits or through physical examination, laboratory test, or other assessments.
Arm/Group | Nivolumab and HF10 (All Participants)
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 3/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab and HF10 (All Participants) (N=7)
Acute kidney injury (Renal and urinary disorders) | 1
Adrenal insufficiency (Endocrine disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 — non-ST-elevation myocardial infarction (NSTEMI), likely demand ischemia
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Endocrine disorders - Other, specify (Endocrine disorders) | 1 — hypophysitis
Esophagitis (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Heart failure (Cardiac disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — basosquamous cell carcinoma
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 — pneumonia left lung
Sepsis (Infections and infestations) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 (2) — lichenoid eruptive keratoacanthomas; squamous cell carcinoma
Thromboembolic event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nivolumab and HF10 (All Participants) (N=7)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1
Chills (General disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Creatinine increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 2 (5)
Dry eye (Eye disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Eye infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 2 (3)
Fatigue (General disorders) | 5 (9)
Flu like symptoms (General disorders) | 5 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Genital edema (Reproductive system and breast disorders) | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1 (3)
Hypothyroidism (Endocrine disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infusion related reaction (General disorders) | 1
Injection site reaction (General disorders) | 2
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Localized edema (General disorders) | 1 (2)
Mucosal infection (Infections and infestations) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — right 3rd digit papule
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — numbness of the lower left ear lobe/jaw
Pain (General disorders) | 1 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Peripheral motor neuropathy (Nervous system disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 (6)
Sinus bradycardia (Cardiac disorders) | 1 (2)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (7) — scalp psoriasis; wasp sting; erythematous plaque; nodular amelanotic area scapha left ear
Skin infection (Infections and infestations) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 1 — shave biopsy of left lateral lower eyelid
Testicular pain (Reproductive system and breast disorders) | 1
Toothache (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-22): https://cdn.clinicaltrials.gov/large-docs/25/NCT03259425/Prot_SAP_003.pdf